CLINICAL TRIAL: NCT05944354
Title: Wearable Spine Health System for Military Readiness
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, William Marras, Principal Investigator, Ohio State University
Other Study IDs: 2022X0054
Record Dates: First submitted 2023-02-06; First posted 2023-07-13 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Low Back Pain; Neck Pain
MeSH Terms: conditions — Low Back Pain; Neck Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Low Back Pain: Subjects with Low Back Pain
- Neck Pain: Subjects with Neck Pain
- Control: Subjects with healthy spines, who have no neck or low back pain
- Operational Air Crew: Subjects that are in training aircrew program

SUMMARY:
The goal of this observational trial is to compare the health history and motion capabilities of participants with low back pain disorders to participants with healthy spines. The main question[s] it aims to answer are to:

1. Primary outcomes of this research effort include the development of composite measures or digital biomarkers to track functional recovery over time and predict duty or work status outcomes (return-to-full duty/work, limited duty/work restrictions or medical discharge/long-term disability).
2. Secondary outcomes of this research effort include characterization of motion assessment utility to predict reinjury risk and evaluate intervention effectiveness. In addition, exploratively, the investigators will determine biopsychosocial profiles of low back pain, and neck pain military populations to identify low back and neck pain phenotypes.

Participants will complete questionnaires and wear a motion monitor that will assess the participant's back and/or neck. This session will be approximately 40-70 minutes. The research team will follow up with participants at 3 month, 6 months, and 1 year to complete a short series of questionnaires and a motion assessment test.

ELIGIBILITY:
Inclusion Criteria:

Control Cohort

* Ages 18-64
* Able to stand for at least 25 minutes
* Able to speak, read, and understand English

Low Back Pain Cohort

* Age 18-64
* Able to stand for at least 15 minutes
* Able to speak, read, and understand English
* Within the last 3 months, an episode of low back pain lasting longer than 7 days and/or seeing a health care provider for low back pain and/or on duty/work restriction due to low back pain.

Neck Pain Cohort

* Ages 18-64
* Able to stand for at least 15 minutes
* Able to speak, read, and understand English
* Within the last 3 months, an episode of neck pain lasting longer than 7 days and/or seeing a health care provider for neck pain and/or on duty/work restriction due to neck pain.

Operational Air crew Cohort

* Ages 18-55
* Able to stand for at least 25 minutes
* Able to speak, read, and understand English
* Ability to participate in cervical and back endurance training programs as part of standard operations

Exclusion Criteria:

Control Cohort

* Known pregnancy
* Within the last 3 months, back or neck pain lasting longer than 7 days and/or seeing a health care provider for low back or neck pain and/or on duty/work restriction due to low back or neck pain.
* Actively being treated by a medical provider for concussion or traumatic brain injury
* Known severe spine curvature or deformity requiring medical treatment (e.g. scoliosis)
* Has been diagnosed by a medical provider with severe vertigo, fainting, narcolepsy, or balance disorders with high risk for falling
* Any known fractures within the last 3 months that will interfere with the motion assessment
* History of spine fracture
* Current condition requiring a bracing or immobilization of the spine
* History of spine surgery (e.g. fusion, micro-discectomy, or artificial disc replacement)
* History of brain or spine cancer
* Currently or within the last 90 days, been treated for cancer with chemotherapy or radiation therapy
* Known severe bone loss or osteoporosis requiring medical treatment and physician-recommended physical restrictions
* Current open wounds on the body where the harnesses will be placed on the neck, head, back, or hips
* Current osteomyelitis or spine infection
* Any other reason that a treating physician, researcher, or participant determines it is unsafe for a patient to perform test

Low Back Pain Cohort

* Known pregnancy
* Current low back pain is the result of a traumatic injury (wreck, fall, etc.) that occurred within the last 3 months OR is positive for spine instability with imaging
* Has spinal fusion across 4 or more lumbar disc levels
* Currently being treated by a medical provider for concussion or traumatic brain injury
* Known severe spine curvature or deformity requiring medical treatment (e.g. scoliosis)
* Has been diagnosed by a medical provider with severe vertigo, fainting, narcolepsy, or balance disorders with high risk for falling
* Any known fractures within the last 3 months that will interfere with the motion assessment
* Any known spinal instability or spine fractures within the last 6 months
* Current condition requiring a bracing or immobilization of the spine
* History of brain or spine cancer
* Currently or within the last 90 days, been treated for cancer with chemotherapy or radiation therapy
* Known severe bone loss or osteoporosis requiring medical treatment and physician-recommended physical restrictions
* Current open wounds on the body where the harnesses will be placed on the back or hips
* Current spine infection or osteomyelitis
* Any other reason that a treating physician, researcher, or participant determines it is unsafe for participant to perform test

Neck Pain Cohort

* Known pregnancy
* Current neck pain is the result of a traumatic injury (wreck, fall, etc.) that occurred within the last 3 months OR is positive for spine instability with imaging
* Has spinal fusion across 4 or more cervical disc levels
* Has an occipital-cervical fusion
* Currently being treated by a medical provider for concussion or traumatic brain injury
* Known severe spine curvature or deformity requiring medical treatment (e.g. scoliosis)
* Has been diagnosed by a medical provider with severe vertigo, fainting, narcolepsy, or balance disorders with high risk for falling
* Any known fractures within the last 3 months that will interfere with the motion assessment
* Any known spinal instability or spine fractures within the last 6 months
* Current condition requiring a bracing or immobilization of the spine
* History of brain or spine cancer
* Currently or within the last 90 days, been treated for cancer with chemotherapy or radiation therapy
* Known severe bone loss or osteoporosis requiring medical treatment and physician-recommended physical restrictions
* Current open wounds on the body where the harnesses will be placed on the neck or head
* Current spine infection or osteomyelitis
* Any other reason that a treating physician, researcher, or participant determines it is unsafe for participant to perform test

Operational Air crew Cohort

* Known pregnancy
* Current neck and/or low back pain is the result of a traumatic injury (wreck, fall, etc.) that occurred within the last 3 months OR is positive for spine instability with imaging
* Has spinal fusion across 4 or more lumbar disc levels
* Currently being treated by a medical provider for concussion or traumatic brain injury
* Known severe spine curvature or deformity requiring medical treatment (e.g. scoliosis)
* Has been diagnosed by a medical provider with severe vertigo, fainting, narcolepsy, or balance disorders with high risk for falling
* Any known fractures within the last 3 months that will interfere with the motion assessment
* Any known spinal instability or spine fractures within the last 6 months
* Current condition requiring a bracing or immobilization of the spine
* History of brain or spine cancer
* Currently or within the last 90 days, been treated for cancer with chemotherapy or radiation therapy
* Known severe bone loss or osteoporosis requiring medical treatment and physician-recommended physical restrictions
* Current open wounds on the body where the harnesses will be placed on the back or hips
* Current spine infection or osteomyelitis
* Any other reason that a treating physician, researcher, or participant determines it is unsafe for participant to perform test

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: There are 4 different study populations: Control, Low Back Pain, Neck Pain, and Operational Air Crew
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Predict Work Status | 2030
  To track functional recovery over time that can predict duty or work status.

SECONDARY OUTCOMES:
Predict Reinjury Risk | 2030
  To track reinjury risk and evaluate intervention effectiveness to predict reinjury risk.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Luke Air Force Base, Luke Air Force Base, Arizona
  - Schriever Space Force Base, Colorado Springs, Colorado
  - Peterson Space Force Base, Colorado Springs, Colorado
  - Eglin Air Force Base, Eglin Air Force Base, Florida
  - Uniformed Services University, Bethesda, Maryland
  - Holloman Air Force Base, Holloman Air Force Base, New Mexico
  - Seymour-Johnson Air Force Base, Seymour-Johnson Air Force Base, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Wright-Patterson Air Force Research Laboratory, Wright-Patterson Air Force Base, Ohio
  - Joint Base Langley- Eustis Air Force Base, Langley Air Force Base, Virginia